CLINICAL TRIAL: NCT07180992
Title: Quantitative and Qualitative Monocytes Analysis and Their Impact on CART Cells Reponse in Multiple Myeloma
Acronym: MONOMM
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0130
Record Dates: First submitted 2025-09-02; First posted 2025-09-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Monocytes; CART Cells
Keywords: Multiple myeloma; Monocytes; CART cells; Microenvironment
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Routine blood withdrawal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tumoral micro-environment in malignant haematological diseases, notably in multiple myeloma, is active on plasma cells survival and proliferation. Monocytosis and monocytes typing are described in multiple myeloma response as factors on proliferation and cell death evasion. CART cells have improved multiple myeloma care in last 5 years, nethertheless, early relapse occur and we must identify predictor factors of better response. The aim of this study is to analyze basic level and phenotyping of monocytes before and after CART cells infusion and study their impact on multiple myeloma response

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Treated for a multiple myeloma
* CART cells treatment proposed
* Affiliated to social security system
* Agreed to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old Treated for a multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
overall response rate | day 1

SECONDARY OUTCOMES:
Progression free survival | 3 years
Overall survival | 3 years
time to next treatment | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No